CLINICAL TRIAL: NCT02266615
Title: Biobank Clinical Genetics Maastricht
Brief Title: Biobank Clinical Genetics Maastricht (KG01)
Acronym: KG01
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC-14-4-077
Record Dates: First submitted 2014-09-18; First posted 2014-10-17 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-05

CONDITIONS: Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA retrieved out of blood or tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Genetic research in 5 areas.: Cardiogenetics; Intellectual Disability, Multiple Congenital Abnormalities and Rare Diseases; Oncogenetics; Dermatogenetics; Reproductive Genetics.
  Interventions: Genetic: Biobanking of biomaterial for future genetic research.

INTERVENTIONS:
Genetic: Biobanking of biomaterial for future genetic research.

SUMMARY:
Collection of coded biomaterial and clinical data with patients consent for future research.

DETAILED DESCRIPTION:
Collection of coded biomaterial and clinical data with patients consent for future research, with the purpose to indentify new gene mutation and prossibilities for treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

* New patients visiting the out patient clinic of the department of Clinical Genetics of the Maastricht University Medical Hospital
* Withdrawal of body material for genetic diagnostics.

Exclusion Criteria:

* Patient does not understand the Dutch language.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New patients visiting the out patient clinic of the department of Clinical Genetics of the Maastricht University Medical Hospital and who get blood or tissue sampled for DNA diagnostics.
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2014-09; Primary Completion 2024-03 (Actual); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Comparing genes to discover unknown functions | Genes will be sequenced and compared, within an expected average of 6 months.
  The biobanked bio material and medical data can be used for future research to learn more about the function of genes.

CONTACTS AND LOCATIONS:
Overall Officials: W. van Zelst-Stams, MD, PhD, Study Director — Head of department
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands